CLINICAL TRIAL: NCT02278198
Title: Evaluation of Thyroid Stunning From a Diagnostic Dose of I-123
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 12-0300
Record Dates: First submitted 2014-10-27; First posted 2014-10-29 (Estimated); Last update posted 2019-10-24 (Actual); Status verified 2019-10

CONDITIONS: Differentiated Thyroid Cancer
Keywords: thyroid cancer
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Thyrotropin Alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Differentiated Thyroid Cancer (Experimental): All patients will receive one extra imaging scan with I-123 in addition to their routine care as described above. This research portion of their care will be similar to the scan that they undergo for the I-123 planning scan that is already a part of their routine care. The research study, which will be performed in the middle of the patient's normal standard of care treatment, will take 4 days.
  On days 1 and 2, all patients will receive a intramuscular injection of rhTSH (Thyrogen).
  On day 3, all patients will be given 3 mCi of I-123 in the form of a pill to take by mouth.
  On day 4, all patients will receive a I-123 Whole Body Imaging Scan and a thyroid camera scan of the neck and thigh.
  Interventions: Drug: rhTSH

INTERVENTIONS:
Drug: rhTSH — Intramuscular injections of rhTSH (Thyrogen) will be given on days 1 and 2.
  Other Names: Thyrogen

SUMMARY:
The purpose of the study is to find out if the small dose of radioiodine, that is used for the dosimetry study on patients with differentiated thyroid cancer, may stun the cancer cells and make the thyroid cancer treatment less effective.

DETAILED DESCRIPTION:
This study plans to learn more about a medical problem called thyroid stunning. Thyroid stunning is a temporary decrease in the function of thyroid cells after small doses of radioiodine, a radioactive drug that is commonly used to treat thyroid cancer. Thyroid stunning can be an important medical problem in patients who have thyroid cancer that has spread beyond the thyroid gland (metastases). In patients with thyroid cancer metastases, some researchers believe it is good to give the maximum safe dose of radioiodine in order to have the greatest chance of destroying the cancer. The maximum safe dose is the highest dose of radioiodine that a patient can safely receive, and this dose is unique to each person. This special personalized dose is determined by first doing a dosimetry study. Dosimetry study is a planning study that calculates the safest dose that the patient can receive. Currently, it is not known whether the small dose of radioiodine that is used for the dosimetry study may stun the cancer cells and make the thyroid cancer treatment less effective.

There are two important types of radioiodine. I-123 is a form of radioiodine that is used to take pictures of the thyroid gland. I-131 is a form of radioiodine that is used to treat thyroid cancer. It is hoped that this study will produce important information that may be the first step in resolving the thyroid stunning question. Investigators will use I-123, a form of iodine that is currently not known to cause thyroid stunning, before thyroid cancer treatment with I-131. Investigators will try to prove that I-123 does not cause thyroid stunning and does not make the thyroid cancer treatment less effective.

Patients are being asked to be in this research study because they have differentiated thyroid cancer, and they have no evidence of thyroid cancer that has spread to the other parts of their body. As a result, those patients thyroid cancer treatment with radioiodine will be a smaller amount than what is needed to treat patients with thyroid cancer that has spread to other parts of the body. Thyroid stunning is not a medical problem for patients like these. However, by participating in this study, the information investigators gather from those patients treatment of thyroid cancer may help those patients with thyroid cancer metastases.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be 21-years-old or greater.
* Patient must be status post near total thyroidectomy for differentiated thyroid cancer without known distant metastases and who are planning to undergo routine remnant thyroid tissue ablation with I-131.
* Patients must qualify for thyroid ablation with I-131.

Exclusion Criteria:

* Women who are pregnant or breastfeeding.
* Prior bovine TSH use.
* Known metastatic thyroid cancer.
* History of cardiovascular disease that may adversely affect patient participation at the discretion of the primary investigator.
* Patients on hemodialysis.
* Patients with acute serious illnesses at the discretion of the primary investigator.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-11-30 (Actual); Primary Completion 2019-09-20 (Actual); Study Completion 2019-09-20 (Actual)

PRIMARY OUTCOMES:
Difference in uptake of I-123 in the thyroid remnant in the neck in the two imaging studies. | 11 days
  Greater than a 20% decrease from the first to second study will indicate evidence of stunning.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Kwak, MD, Principal Investigator — Department of Radiology
Locations (1):
- Fawn N White, Denver, Colorado, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-26): https://cdn.clinicaltrials.gov/large-docs/98/NCT02278198/Prot_SAP_000.pdf